CLINICAL TRIAL: NCT04422535
Title: Observational Study to Evaluate the Effects on the Qt Interval of COVID-19 Coronavirus Infection in Critically Ill Patients
Brief Title: Effects on the Qt Interval of COVID-19 Coronavirus Infection
Acronym: QT-COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Matilde Zaballos (Other)
Responsible Party: Sponsor-Investigator, Matilde Zaballos, specialist physician at Anesthesiology Department, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: QT-COVID-19
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus Infection; Intensive Care Patients
Keywords: QT interval, ventricular repolarization
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical care patients: Patients admitted to critical care units for COVID-19, where ECG records and relevant clinical information are available to assess the impact of the disease and its concomitant treatment on electrocardiographic parameters of ventricular repolarization

SUMMARY:
The present study aims to evaluate the impact of COVID-19 disease and its treatment on ventricular repolarization, assessed by measuring the QTc interval, in patients admitted to the critical care unit.

DETAILED DESCRIPTION:
Coronavirus infection of Severe Acute Respiratory Syndrome COVID-2 is characterized by a broad clinical spectrum ranging from asymptomatic infection, mild upper respiratory tract disease and severe viral pneumonia with respiratory failure and even death, with many patients hospitalized with pneumonia. In addition, the infection can have a direct impact on cardiovascular disease including the development of arrhythmias, although the exact incidence is not known. Treatments administered for COVID-19 infection have the potential to produce adverse cardiovascular effects including prolongation of the QT interval and development of arrhythmias.

Relevant clinical data that may affect the QT interval and specifically the medication the patient has received will be recorded. The specific treatment administered for COVID-19 will be recorded as the concomitant medication of the critical patient that may have an impact on the QT interval. Analytical data will also be collected on plasma levels of ions such as potassium, calcium and magnesium, blood gases, renal and hepatic function parameters and cardiac markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to intensive care units for COVID-19 infection with an ECG record

Exclusion Criteria:

* Patients in critical care unit without COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients admitted to critical care units with COVID-19 infection
  * Ages between 18-80 years
  * Documentation in the clinical history sufficient to collect the data of interest to the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the QT and QTc interval in patients admitted to intensive care units for COVID-19 infection | through study completion, an average of 1 year
  The QT interval measurement will be performed on the available 12-lead ECG from the medical record. The QT interval will be measured according to the recommendations of the scientific societies of cardiology: it is considered from the beginning of the activation of the ventricular myocardium and the end of its repolarization, which are represented in the ECG respectively by the beginning of the QRS and the end of the T wave. Ideally, the QT interval should be measured in Q-wave leads in DII and V5. An average value of 3 heart cycles (beats) should be recorded. Two researchers to control inter-observer variability will perform the measurement.

SECONDARY OUTCOMES:
incidence of arrhythmias and impact of the COVI-drugs administered on QT interval | through study completion, an average of 1 year
  To assess the incidence of arrhythmias in critically ill patients with COVID-19 infection admitted to critical patient units.
  To evaluate the impact of the association of drugs administered for the treatment of COVID-19 infection in critically ill patients in the QT interval.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Hortal, MD PhD, Study Chair — Hospital Universitario Gregorio Marañon
Locations (1):
- Servicio de Anestesia, Hospital General Universitario Gregorio Marañon, Madrid, Spain

REFERENCES:
- [Result] Fernandes FM, Silva EP, Martins RR, Oliveira AG. QTc interval prolongation in critically ill patients: Prevalence, risk factors and associated medications. PLoS One. 2018 Jun 13;13(6):e0199028. doi: 10.1371/journal.pone.0199028. eCollection 2018. PMID 29898002
- [Result] Pickham D, Helfenbein E, Shinn JA, Chan G, Funk M, Drew BJ. How many patients need QT interval monitoring in critical care units? Preliminary report of the QT in Practice study. J Electrocardiol. 2010 Nov-Dec;43(6):572-6. doi: 10.1016/j.jelectrocard.2010.05.016. PMID 21040827
- [Result] Gowda RM, Khan IA, Wilbur SL, Vasavada BC, Sacchi TJ. Torsade de pointes: the clinical considerations. Int J Cardiol. 2004 Jul;96(1):1-6. doi: 10.1016/j.ijcard.2003.04.055. PMID 15203254
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816